CLINICAL TRIAL: NCT04245293
Title: Open, Comparative Study To Evaluate The Performance And Safety Of The Medical Device AINARA® Vaginal Gel Versus A Hyaluronic Acid-Based Gel In Late Menopausal Transition Women Affected By Vaginal Dryness
Brief Title: Clinical Trial Study To Evaluate The Performance And Safety Of Ainara®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Italfarmaco (Industry)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DMS/18/AINARA/01
Record Dates: First submitted 2020-01-27; First posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Vaginal Disease
MeSH Terms: conditions — Vaginal Diseases

STUDY DESIGN:
Intervention Model Description: This is an open-label, comparative, multicenter study with two parallel group of subjects. The clinical investigation will be performed in three clinical sites.
  The calculated sample size of subjects is 50 (25 subject for each arm). To obtain this number of evaluable subjects it will be needed to screen about 60 subjects (including 6 potential screening failure) and to enroll 54 subjects (estimating 4 subjects drop out). From the equal distribution per groups of treatment point of view, the minimum and maximum number of patients recommended for each of the three centers will be 8 and 25, respectively.
  The research question is: in a population of menopausal transition women affected by vaginal dryness, will a 1-month treatment with polycarbophilic vaginal gel (Ainara®) significantly decrease the symptomatology evaluated by VHI and VAS in comparison with that occurred in a group of patients treated with a HA-based gel (HyaloGyn®)?
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ainara (Experimental): Experimental: Ainara Each administration kit (subject kit) for patients of Ainara® will contain a box with 1 tube with 30 g gel, 1 cannula and 1 plunger. The gel quantity is enough for one subject over the course of the study (1 g at each administration).
  Interventions: Device: Ainara
- HyaloGin (Active Comparator): Active Comparator: HyaloGin Each administration kit (subject kit) for patients allocated to HyaloGyn® group will contain a box with: 1 tube with 30g gel and 10 single-use applicators consisting of a piston and one opaque plastic plunger.
  The gel quantity is enough for one subject (3g application every three days over the course of the study).
  Interventions: Device: HyaloGin

INTERVENTIONS:
Device: Ainara — Each administration kit (subject kit) for patients of Ainara® will contain a box with 1 tube with 30 g gel, 1 cannula and 1 plunger. The gel quantity is enough for one subject over the course of the study (1 g at each administration).
  Arms: Ainara
Device: HyaloGin — Active Comparator: HyaloGin Each administration kit (subject kit) for patients allocated to HyaloGyn® group will contain a box with: 1 tube with 30g gel and 10 single-use applicators consisting of a piston and one opaque plastic plunger.
  The gel quantity is enough for one subject (3g application every three days over the course of the study).
  Arms: HyaloGin

SUMMARY:
This study evaluates treatment with the medical device Ainara® compared to a HA-based gel (Hyalogin) on the improvement of vaginal dryness

DETAILED DESCRIPTION:
This is an open, comparative, multicenter study that evaluates the performance and safety of the medical device Ainara®.

In this study we use polycarbophilic vaginal moisturizing gel (Ainara®) compared with a HA-based gel (Hyalogin) for symptomatic treatment of vaginal dryness and we will monitor its impact on vaginal dryness symptoms evaluated by Vaginal Health Index and Vaginal Analogue Scale.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant and in menopausal transition period (late peri-menopause) women following the STRAW criteria and with a break in menstrual periods of at least 60 days, aged ≥ 45 to ≤ 55 years.
* Diagnosis of vaginal dryness by subjective dryness, any objective sign of VVA, pH>5 as reported in the AGATA study and VHI < 15.
* Body mass index of ≥ 18.5 to ≤ 36 kg/m2.
* Females of child bearing potential who agree to use only lubricated condoms or spiral as contraceptives methods, during the full duration of the study.
* Able to communicate adequately with the Investigator and to comply with the requirements for the entire study.
* Capable of and freely willing to provide written informed consent prior to participating in the study.

Exclusion Criteria:

* Women in post-menopausal (total cessation of menses for ≥ 1 year from the date of the screening visit).
* Malignancy (also leukemic infiltrates) within 5 years prior to day 0 (except for treated basal cell/squamous cell carcinoma of the skin).
* Genital bleeding.
* Estrogen vaginal treatment during the study period (permitted only if terminated at least 6 months before study).
* Systemic estrogen therapy (permitted only if terminated at least 6 months before study).
* Subjects with illness, or other medical condition that, in the opinion of the investigator, would compromise participation or be likely to lead to hospitalization during the course of the study.
* Clinical evidence of acute infection currently requiring treatment (syphilis, herpes simplex, human papilloma virus, gonorrhoea, chlamydia, lymphogranuloma venereum, etc.); clinical evidence or history of chronic infectious disease (i.e. tuberculosis).
* Psychosis, schizophrenia, mania, depressive disorders, history of suicide attempt or suicidal ideation, or any other psychiatric illness (except for intermittent anxiety).
* Known allergy to tested IMDs or its excipients.
* Drug or alcohol abuse within 12 months of Day 0.
* Participation in an interventional clinical study or administration of any investigational agents in the previous 30 days.
* Presence of any clinically significant medical condition judged by the investigator to preclude the patient's inclusion in the study

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
The Vaginal Health Index (VHI) | 30 days
  The changing from baseline to day 30 (final visit) for VHI mean value in each group separately and the changing in the Ainara® group in comparison with that occurred in HyaloGyn® group; The minim score is 5 and the maxim is is 25
Visual Analogue Scale (VAS) | 30 days
  The changing from baseline to day 3, 7, 21, 30 (final visit) for VAS mean value in each group separately and in the Ainara® group in comparison with that occurred in HyaloGyn® group. The minim score is 0 and the maxim score is 5, where 0 represents no symptoms and 3 represents severe symptoms

SECONDARY OUTCOMES:
subjective symptoms | 30 days
  Subjective symptoms dryness, itching, burning, dyspareunia, and dysuria reported on patient diary and scored as reported in the AGATA study as follows:
  0 = absence, 1 = slight, 2 = moderate, and 3 = severe intensity. The change in these variables will be evaluated from baseline to day 3, 7, 21, 30 (final visit).
objective signs in the vaginal mucosa | 30 days
  Objective signs in the vaginal mucosa: dryness, thinning rugae, pallor, fragility, and petechiae scored as reported in the AGATA study as follows:
  0 = absence, 1 = slight, 2 = moderate, and 3 = severe alteration. For these variables will be evaluated the changing from baseline to day 3, 7, 21, 30 (final visit) with comparison intra and inter groups.
Vaginal pH | 30 days
  It will be measured by the Investigators with a test strip delivered by Sponsor. The baseline values can be from 5.0 (this was the minimum value need for vaginal atrophy diagnosis in AGATA study) to 9.0. The Investigator will insert the pH strip into the upper wall of the vagina and will consider the reading made while the strip is still damp. For this outcome will be analysed the changing of mean values from baseline to 30 day (final visit) with comparison intra and inter groups.
Vaginal Trophism Maturation Value (MV) | 30 days
  Vaginal Trophism Maturation Value (MV): this outcome will be obtained from the cellular count of the vaginal smears at baseline and at the 30 days visit. The samples will be fixed, stored, and sent in the local laboratory in Timisoara, Romania (address details in TMF) for staining (Papanicolaou technique) and subsequent analysis. Samples will be evaluated by one independent cytopathologist blinded to the treatment. The MV will be calculated according to the following: MV = [1x (% superficial cells)] + [0.6x (% intermediate cells)] + [0.2x (% parabasal cells)]. The comparison intra and inter groups will be between baseline values and 30 days values.
Female Sexual Function Index (FSFI) | 30 days
  Female Sexual Function Index (FSFI) Romanian version, evaluated by Investigator and analysed considering the changing from baseline to 30 days (final visit) with comparison intra and inter groups.
Sexual Function (SF 12) | 30 days
  SF 12 (Romanian version) evaluated by Investigator and analysed considering the changing from baseline to 30 day (final visit) with comparison intra and inter groups.
Global Symptom Score (GSS) | 30 days
  Global Symptom Score (GSS) a composite score of symptoms, will be obtained to assess the effect of treatment on all individual symptoms taken as a whole. It will be calculated by the addition of the intensity scores of all individual symptoms (range, 1-15: 1 = only mild vaginal dryness, 15 = all five symptoms severe in intensity). This outcome will be compared intra and inter groups, assessing the changing from baseline visit to 30 days visit (final visit).
Patient Global Assessment of Safety (PGAS) | 30 days
  Patient Global Assessment of Safety (PGAS): it will be reported by the subject at all visits and all phone contacts in the patient diary using the 4-point scale:
  1= very good safety, 2 = good safety, 3 = moderate safety and 4 = poor safety.
Investigator Global Assessment of Safety (IGAS) | 30 days
  Investigator Global Assessment of Safety (IGAS): it will be reported by the Investigator using the 4-point scale:
  1= very good safety, 2 = good safety, 3 = moderate safety and 4 = poor safety. IGAS will be evaluated at the last visit, only.
Adverse Event, Adverse Device Event, Serious Adverse Event, Suspected Adverse Device Event | 30 days
  AE, ADE, SAE, SADE: they will be reported by the Investigators according to the current legislation. All adverse events will be collected by Investigators at all visits and phone contacts and evaluated considering the change from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Liviu Cristian PĂTRAȘCU, Dr, Principal Investigator — Fizio Center
Locations (1):
- Fizio Center, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: No